CLINICAL TRIAL: NCT02848833
Title: A Regulatory Requirement Non Interventional Study to Monitor the Safety and Effectiveness of JARDIANCE® (Empagliflozin, 10mg, 25mg, q.d.) in Korean Patients With Type 2 Diabetes Mellitus
Brief Title: JARDIANCE Regulartory Post Marketing Surveillance in Korean Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245.116
Record Dates: First submitted 2016-06-27; First posted 2016-07-29 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- JARDIANCE: T2DM with JARDIANCE
  Interventions: Drug: JARDIANCE 10mg; Drug: JARDIANCE 25mg

INTERVENTIONS:
Drug: JARDIANCE 10mg — T2DM with JARDIANCE 10mg
Drug: JARDIANCE 25mg — MT2DM with JARDIANCE 25mgax

SUMMARY:
To monitor the safety profile and effectiveness of Empagliflozin in Korea patients with type 2 diabetes mellitus in a routine clinical practice setting

ELIGIBILITY:
Inclusion criteria:

1. Patients who have been started on JARDIANCE® in accordance with the approved label in Korea
2. Age = 19 years at enrolment
3. Patients who have signed on the data release consent form

Exclusion criteria:

1. Known hypersensitivity to empagliflozin or any of its excipients
2. Patients with type 1 diabetes or for the treatment of diabetic ketoacidosis
3. Patients with persistent estimated Glomerular Filtration Rate <60 mL/min/1.73 m2,end stage renal disease or on dialysis
4. Patients with rare hereditary conditions of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
5. Patients for whom empagliflozin is contraindicated according local label of JARDIANCE®

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes mellitus in Korea
Sampling Method: Probability Sample
Enrollment: 3368 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, South Korea

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was and observational prospective, non-interventional, open-label, multi-centre study to monitor the safety profile and efficacy of JARDIANCE® (empagliflozin, 10 milligram (mg), 25mg) in Korean patients with type 2 diabetes mellitus in a routine clinical practice setting.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- JARDIANCE®: JARDIANCE® was prescribed according to the local label and at the discretion of the treating physician. The recommended dose of JARDIANCE® was 10 milligram (mg) once daily. In patients tolerating JARDIANCE® 10 mg once daily and requiring additional glycemic control, the dose could be increased to 25 mg once daily. When JARDIANCE® was used in combination with a sulphonylurea or with insulin, a lower dose of the sulphonylurea or insulin was considered to reduce the risk of hypoglycaemia. JARDIANCE® could be taken with or without food and tablets and was swallowed whole. If a dose was missed, it was taken as soon as the patient remembered. A double dose was not taken on the same day.
Period: Overall Study
Arm/Group | JARDIANCE®
Started | 3368
Completed (All Participants whose case report forms (CRFs) were retrieved during the re-examination period and who did not violate the inclusion/exclusion criteria.) | 3231
Not Completed | 137
Not completed — subject who are duplicated | 1
Not completed — have not taken the study drug | 11
Not completed — follow-up failure | 6
Not completed — Protocol Violation | 119

BASELINE CHARACTERISTICS:
Population: Safety analysis set: All Participants who signed the informed consent form to participate in this study as subject, took JARDIANCE® once at least, and were followed up by the physician once or more.
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 3231
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.66 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1380
  Male | 1851
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Events
Description: Percentage of participants with any adverse events was reported. The 95% Confidence Interval for the percentage of participants with adverse events was calculated by Exact Method.
Time Frame: From baseline (Visit 1) until last visit (the last follow-up visit a patient actually attended during the study), up to 544 days.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 3231
Percentage of participants | 13.93 [12.75 to 15.17]

2. Primary Outcome: Percentage of Participants With Adverse Events Relating to Study Drug
Description: Percentage of participants with adverse events relating to study drug was reported. The 95% Confidence Interval for the percentage of participants with adverse events was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 3231
Percentage of participants | 5.14 [4.40 to 5.96]

3. Primary Outcome: Percentage of Participants With Unexpected Adverse Events
Description: Percentage of participants with unexpected adverse events was reported. The 95% Confidence Interval for the percentage of participants with adverse events was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 3231
Percentage of participants | 11.54 [10.46 to 12.70]

4. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest
Description: Percentage of participants with adverse events of special interest (AESI) was reported. The 95% Confidence Interval for the percentage of participants with adverse events was calculated by Exact Method.
  The following are considered as AESIs:
  * Vaginal moniliasis, vulvovaginitis, balanitis and other genital infection
  * Increased urination
  * Urinary tract infection (UTI)
  * Volume depletion
  * Diabetic Ketoacidosis (DKA)
  * Decreased renal function:
  * Hepatic injury
  * Lower limb amputation
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 3231
Percentage of participants | 1.45 [1.07 to 1.93]

5. Primary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation of the Drug
Description: Percentage of participants with adverse events leading to discontinuation of the drug was reported. The 95% Confidence Interval for the percentage of participants with adverse events was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 3231
Percentage of participants | 3.25 [2.67 to 3.92]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Last Visit
Description: Change from baseline in glycosylated hemoglobin (HbA1c) at last visit.
Time Frame: At baseline (Visit 1) and at the last visit (the last follow-up visit a patient actually attended during the study, up to day 544).
Population: Effectiveness analysis set: All Participants who signed the informed consent form to participate in this study as subject, visited as per the study schedule, took JARDIANCE®, and were evaluated for the efficacy.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2567
Percentage of glycosylated hemoglobin | -0.68 (1.39)
Statistical Analysis 1: Comparison: JARDIANCE®; Test type: Other; p < 0.0001, paired t-test — Difference before administration versus after administration was analyzed using a paired t-test

7. Secondary Outcome: Number of Patients Who Had Glycosylated Hemoglobin (HbA1c) Reaching Less Than 7% (Target Efficacy Response Rate) at the Last Visit
Description: Number of patients who had glycosylated hemoglobin (HbA1c) reaching less than 7% (target efficacy response rate) at the last visit.
Time Frame: At the last visit (the last follow-up visit a patient actually attended during the study, up to day 544).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2567
Participants
  lower than 7% | 1132
  greater than or equal to 7% | 1435

8. Secondary Outcome: Number of Patients With Relative Effectiveness Response in Glycosylated Hemoglobin (HbA1c) (Decrease by at Least 0.5% Comparing to Baseline) at the Last Visit
Description: Number of patients with relative effectiveness response in glycosylated hemoglobin (HbA1c) (decrease by at least 0.5% comparing to baseline) at the last visit
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2567
Participants
  greater than or equal to 0.5% | 1315
  lower than 0.5% | 1252

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Last Visit
Description: Change from baseline in fasting plasma glucose (FPG) at last visit.
Time Frame: as for outcome 6
Population: Effectiveness analysis set: All Participants who signed the informed consent form to participate in this study as subject, visited as per the study schedule, took JARDIANCE®, and were evaluated for the efficacy. Only those subjects with non-missing outcome measures were included in this analysis.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dl)
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2160
milligram per deciliter (mg/dl) | -25.59 (59.84)
Statistical Analysis 1: Comparison: JARDIANCE®; Test type: Other; p < 0.0001, paired t-test — Difference before administration versus after administration was analyzed using a paired t-test

10. Secondary Outcome: Change From Baseline in Body Weight at Last Visit
Description: Change from baseline in body weight at last visit.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2097
kilogram | -1.91 (3.37)
Statistical Analysis 1: Comparison: JARDIANCE®; Test type: Other — Difference before administration versus after administration was analyzed using a paired t-test; p < 0.0001, paired t-test

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Last Visit
Description: Change from baseline in systolic blood pressure (SBP) at last visit.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2355
millimeters of mercury (mmHg) | -3.95 (15.44)
Statistical Analysis 1: Comparison: JARDIANCE®; Test type: Other; p < 0.0001, paired t-test — Difference before administration versus after administration was analyzed using a paired t-test

12. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Last Visit
Description: Change from baseline in diastolic blood pressure (DBP) at last visit.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2354
millimeters of mercury (mmHg) | -1.80 (10.82)
Statistical Analysis 1: Comparison: JARDIANCE®; Test type: Other; p < 0.0001, paired t-test — Difference before administration versus after administration was analyzed using a paired t-test

13. Secondary Outcome: Number of Participants Per Final Effectiveness Assessment Category at Last Visit
Description: Number of participants per final effectiveness assessment category at last visit was reported. The final effeciveness consisted of 4 categories: Improved (If determined as there was any effect of maintaining or improving disease related factors.), Unchanged (If disease related factors had not been changed compared with before administration, and not determined as there was any effect of maintaining symptoms.), Aggravated (If disease related factors were worse than before administration.), and Unassessable (If it cannot be determined due to insufficient information collected.).
Time Frame: At the last visit (the last follow-up visit a patient actually attended during the study, up to day 544).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 2567
Participants
  Improved | 1749
  Unchanged | 546
  Aggravated | 195
  Unassessable | 77

ADVERSE EVENTS:
Time Frame: From baseline (Visit 1) until last visit (the last follow-up visit a patient actually attended during the study), up to 544 days.
Description: Safety analysis set: All Participants who signed the informed consent form to participate in this study as subject, took JARDIANCE® once at least, and were followed up by the physician once or more.
Arm/Group | JARDIANCE®
All-Cause Mortality (participants affected / at risk) | 0/3231
Serious Adverse Events (participants affected / at risk) | 55/3231
Other Adverse Events (participants affected / at risk) | 0/3231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JARDIANCE® (N=3231)
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 4
Coronary artery disease (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 2
Glaucoma (Eye disorders) | 1
Pathologic myopia (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Rhegmatogenous retinal detachment (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Vascular stent stenosis (General disorders) | 1
Vascular stent thrombosis (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendiceal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tubo-ovarian abscess (Infections and infestations) | 1
Vestibular neuronitis (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Splenic injury (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Cervix inflammation (Reproductive system and breast disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Benign neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02848833/Prot_SAP_000.pdf